CLINICAL TRIAL: NCT06072859
Title: The Impact of Simulated Forest Immersion Therapy on Pain and Anxiety in Patients Axial Spondyloarthritis (axSpA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Amy Ross, Associate Professor, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 00025267
Record Dates: First submitted 2023-09-26; First posted 2023-10-10 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Axial Spondyloarthritis
Keywords: Forest Oils; Volatile Organic Compounds; Terpenes; Virtual Reality; Pain; Anxiety; Mood
MeSH Terms: conditions — Axial Spondyloarthritis; Pain; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Feasibility quasi-experimental
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator): Humidified Forest Oils with Limonene
  Interventions: Other: Humidified Forest Oils
- Group 2 (Active Comparator): Forest oils and audio-visual forest exposure
  Interventions: Other: Forest oils and audio-visual forest exposure

INTERVENTIONS:
Other: Humidified Forest Oils — 60mls Limonene in 200mls water humidified with a diffuser.
  Arms: Group 1
Other: Forest oils and audio-visual forest exposure — 60mls Limonene in 200mls water humidified with a diffuser and audiovisual Forest sights and sounds on Surface Pro tablet.
  Arms: Group 2

SUMMARY:
The purpose of the study is to learn about the ease of using a humidified fragrant citrus forest oil, along with a virtual simulation of a forest environment (i.e., with sights and sounds of nature using a personal tablet Surface Pro 3 with headphones, to learn more about how these two aspects of the simulated forest immersion therapy (SFIT) may improve pain, anxiety, blood-pressure, and heart rate related to Axial Spondyloarthritis. The investigators hope to learn how well SFIT may impact pain levels, feelings of calm, as well as blood- pressure and heart rate, and how participants tolerate the experience overall.

DETAILED DESCRIPTION:
DURATION:

Participation in the study will consist of 1 visit total and will last up to 2 consecutive hours.

PROCEDURES:

Participants will be randomized to receive either the forest oils only, or the forest oils and audio-visual forest exposure described above for up to 1 hour.

Study Visit:

* During Visit 1 and the only study visit, the investigator will explain the study and obtain consent. The Investigator will explain this study and answer any questions the participant may have. The participant will have the opportunity to review this document in detail.
* Consent may be withdrawn by the participant at any time during the study.
* Once the written consent is signed, the participant will be asked to rest for 15 minutes.
* During the resting period, randomization will occur into one of two groups:
* Group 1 - Forest oils only, or
* Group 2 - Forest oils and audio-visual forest exposure
* Following the resting period, demographics will be collected from the participants.
* The investigators will then take a blood pressure and heart rate measurement.
* Then, the investigator will ask the participants to fill out two questionnaires. One of these questionnaires consists of two questions asking the participants about their pain level and location, the other questionnaire asks about mood state and how the participants rate various qualities of their feelings. The third questionnaire asks the participants about their pain levels specific to the past week.
* Participants will then be taken into the study room where they will participate in the simulated forest experience.
* If the participants are randomly assigned to Group 1, they will be breathing in the aroma of the forest oils for a period of 1 hour in the study room. There is an adjustable lounge chair in the room to sit in. And the participants may read or use their phone quietly.
* If the participants are randomly assigned to Group 2, they will be breathing in the aroma of the forest oils for a period of 1 hour in the study room while using the headphones and tablet with the simulated forest greenspace sights and sounds. There is an adjustable lounge chair in the room to sit in.
* The investigator will take the participants blood pressure and heart rate measurement after 30 minutes from the start of the intervention.
* Within 15 minutes following the simulated experience in the study room, the investigator will take one more blood-pressure and heart rate measurement. Then, the participants will fill out the same two questionnaires again, which are asking the participants about their pain level and location and mood.
* The investigators will then ask the participants some questions about the participants' experience before the end of the study visit.
* One week after the participants study visit (Study Visit 1), the investigator will ask the participants to return two follow-up questionnaires to us over encrypted and password protected OHSU email, or by arranging to drop the questionnaires off with the Study Coordinator or the Rheumatology Clinic at OHSU.

RISKS: There are three risks to participation in this study and these are all considered minimal risks. Participants may have an allergic reaction, a cough, or an increase in asthma type symptoms, such as difficulty breathing related to the humidified fragrant citrus forest oil used in this study. For those in Group 2, the participants may experience a sensation of nausea (feeling queasy), discomfort related to the headphone placement, sound disturbances related to the volume of the nature sounds, or discomfort related to viewing the images of the forest greenspace environment utilized in this study. the investigators will make every effort to protect the participants privacy during this study, including password protected files, secure and encrypted email, and double locked file system. A loss of confidentiality happens when the participants private information is accessed outside the scope of this study. A loss of confidentiality is an unexpected event.

BENEFITS: Participants may not directly benefit from taking part in this research. However, participation will potentially benefit patients with Axial Spondyloarthritis in the future.

ELIGIBILITY:
Inclusion Criteria:

* able to read at a 5th grad level
* medically diagnosed with Axial Spondyloarthritis
* tolerate having their BP and HR taken
* average of greater than 3 on their last recorded pain assessments
* average of greater than 4 on their last BASDI recorded
* currently have an assigned Rheumatologist in their care delivery

Exclusion Criteria:

* history of asthma
* currently pregnant
* inability to detect common odors from commercial fragrances
* smoking within 15 minutes of the start of the intervention procedure
* known allergy to citrus aroma
* hard of hearing without assistive devices
* limited vision not corrected by eye lenses
* history of hypertension uncontrolled by medications

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-09-21 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Axial Skeleton Pain | before intervention on visit 1, directly after intervention on visit 1, and one week later
  Pain on Visual Analog Scale, Scores 0-10 with higher scores reflecting greater pain
Anxiety | before intervention on visit 1, directly after intervention on visit 1, and one week later
  Anxiety as scored on STAI - State only Higher scores mean greater state anxiety, 20 items with a scoring range of 1-4 on each of them. Score is totaled and range 20-80 with higher scores reflecting higher anxiety as a state.
Blood Pressure | before intervention on visit 1, after 30 minutes of the intervention start on visit 1, directly after intervention on visit 1, and one week later
  Blood Pressure measured by Omnicron tabletop BP and HR device, used clinically, higher Blood Pressure, both systolic and diastolic pressures, measured reflect/correlate with higher anxiety or pain status. Measure range 0-240.
Heart Rate | before intervention on visit 1, after 30 minutes of the intervention start on visit 1, directly after intervention on visit 1, and one week later
  Heart Rate measured by Omnicron tabletop BP and HR device, used clinically, higher Heart Rate measured reflect/correlate with higher anxiety or pain status. Measure range 0-300.
Feasibility Questions | directly after intervention on visit 1
  Questions regarding the intervention include the tolerance of the intervention, likes and dislikes of the experience and any suggestions to make the intervention experience better.

SECONDARY OUTCOMES:
Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) | before intervention on visit 1, directly after intervention on visit 1, and one week later
  Measures pain and functionality in Axial Spondyloarthritis by assessing individual metrics for fatigue, axial involvement, peripheral articular involvement, localized tenderness/enthesitis, and morning stiffness. Score 0-10 with higher scores reflecting higher pain and functionality issues.
Routine Assessment of Patient Index Data 3 (RAPID3) | before intervention on visit 1, directly after intervention on visit 1, and one week later
  composite index which is routinely and reliably used to assess disease activity in Axial Spondyloarthritis. Score range 0-30 with higher scores reflecting higher disease activity.

CONTACTS AND LOCATIONS:
Overall Officials: Amy Miner Ross, PhD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No